CLINICAL TRIAL: NCT03997292
Title: Intravenous ThrombolysisRegistry for Acute Ischemic Stroke in China
Brief Title: Intravenous Thrombolysis Registry for Acute Ischemic Stroke in China
Status: Withdrawn | Type: Observational
Why Stopped: The study has been terminated due to key change of protocol
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Neurology Chief, General Hospital of Shenyang Military Region
Other Study IDs: K201707
Record Dates: First submitted 2017-11-14; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Ischemic Stroke
Keywords: alteplase; urokinase; intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator; Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Alteplase group: According to 0.6-0.9mg / kg alteplase (maximum can not exceed 90mg), of which 10% intravenous injection, the remaining 60 minutes intravenous infusion
  Interventions: Drug: Alteplase
- Urokinase group: 1.2-1.5 million U dissolved in 100ml sodium chloride injection, 30 minutes intravenously End
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Alteplase — According to 0.6-0.9mg / kg alteplase (maximum can not exceed 90mg), of which 10% intravenous injection, the remaining 60 minutes intravenous infusion.
  Groups: Alteplase group
Drug: Urokinase — 1.2-1.5 million U dissolved in 100ml sodium chloride injection, 30 minutes intravenously.
  Groups: Urokinase group

SUMMARY:
To analyze the real situation of intravenous thrombolysis in acute ischemic stroke in China

DETAILED DESCRIPTION:
Compare the efficacy and safety of different thrombolytic drugs; Analysis of patients during hospital treatment of adverse events and complications; Analysis of factors that affect the effectiveness of treatment; Evaluate the pharmacological benefits of different thrombolytic drugs

ELIGIBILITY:
Inclusion Criteria:

* 1) age> 18 years old;
* 2) meet the diagnostic criteria of China 2014 guidelines for the diagnosis and treatment of acute ischemic stroke;
* 3) no history of first sepsis or previous cerebral infarction sequelae (mRS ≤ 1);
* 4) within 3 hours of onset;
* 5) Have measurable neurological deficits;
* 6) Patients or legal guardians can understand and sign informed consent.

Exclusion Criteria:

* Absolute exclusion criteria:
* 1) history of head trauma or stroke within the last 3 months;
* 2) suspected subarachnoid hemorrhage;
* 3) history of previous intracranial hemorrhage;
* 4) intracranial tumor, arteriovenous malformation or aneurysm ;
* 5) recent intracranial or intraspinal surgery;
* 6) arterial puncture at an incurable site within the last 7 days;
* 7) elevated blood pressure: systolic blood pressure ≥180 mm Hg, or diastolic blood pressure ≥100 mm Hg;
* 8) Internal bleeding;
* 9) acute bleeding tendency, including platelet count less than 100 × 109 / L or other conditions;
* 10) heparin treatment within 48 h (APTT is outside the upper limit of normal range);
* 11) oral anticoagulant, INR> 1.7 Or PT> 15S;
* 12) are currently using thrombin inhibitors or factor Xa inhibitors, various sensitive laboratory abnormalities (such as APTT, INR, platelet count, ECT; TT or appropriate factor Xa activity assays) ;
* 13) Blood glucose <50 mg / dl (2.7 mmol / L);
* 14) CT suggestive of multiple cerebral infarction (low density range> 1/3 of the cerebral hemispheres) ;
* 15) Other conditions considered unsuitable for inclusion in this clinical study;
* 16) 3 months or are participating in other clinical trials;
* 17) combined with severe systemic disease is expected to survive less than three months.
* Relative exclusion criteria:
* 1) severe stroke (NIHSS> 25 points);
* 2) pregnancy;
* 3) neurological deficits after epileptic seizures;
* 4) major surgery or severe trauma within the last 14 days;
* 5) Urethral hemorrhage;
* 6) Myocardial infarction within the last 3 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thrombolytic patients with acute ischemic stroke within 3 hours of onset
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
mRS of 90 days after thrombolysis | Month 3
  Proportion of patients with mRS = 0-1 points 90 days after thrombolysis

SECONDARY OUTCOMES:
Evaluation of Adverse events | Year 1
  Symptomatic intracranial hemorrhage conversion rate; Liver and kidney dysfunction; Bleeding gums; Skin mucous membrane bleeding

OTHER OUTCOMES:
Economic evaluation | Day 14
  The cost-effectiveness of different thrombolytic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, doctor, Principal Investigator — Neurology Chief
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided